CLINICAL TRIAL: NCT02414698
Title: Single Center, Randomized PROspective Study Comparing Percutaneous HydroDiscectomy to Transforaminal Epidural Steroid Injections in the Treatment Of Radiculopathy Secondary to Lumbar Disc Herniation (PROPHESOR)
Brief Title: Percutaneous HydroDiscectomy Compared to TESI for Radiculopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Integral investigator left study; could not continue recruiting.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-3750
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Hydrodiscectomy (Active Comparator): Percutaneous Hydrodiscectomy with the SpineJet Hydrodiscectomy System
  Interventions: Procedure: Percutaneous Hydrodiscectomy
- TESI (Active Comparator): Transforaminal Epidural Steroid Injections
  Interventions: Drug: TESI

INTERVENTIONS:
Procedure: Percutaneous Hydrodiscectomy — The HydroD uses a thin supersonic stream of water to cut, ablation, remove disc material percutaneously via a skin puncture.
  Arms: Percutaneous Hydrodiscectomy
Drug: TESI — Transforaminal epidural steroid injections given in the lumbar spine.
  Other Names: Transforaminal epidural steroid injections
  Arms: TESI

SUMMARY:
To compare the outcomes of percutaneous lumbar Hydrodiscectomy (HydroD) with the SpineJet Hydrodiscectomy System to transforaminal epidural steroid injections (TESI) in patients with lumbar radiculopathy due to contained disc herniation with symptoms that persist following a treatment course of conservative management including physical therapy and anti-inflammatory medication.

DETAILED DESCRIPTION:
Lumbar disc herniation is one of the leading causes of lower back pain and sciatica. If conservative management fails to relieve radiculopathy secondary to lumbar disc herniation, interventional treatments such as epidural steroid injections are indicated. Patients that do not have pain relief from transforaminal epidural steroid injections or over time relief is diminished, surgical intervention is typically recommended and microdiscectomy is the surgical intervention of choice. Over the years, a number of minimally invasive techniques for lumbar disc herniation have been introduced including percutaneous mechanical lumbar discectomy, including percutaneous hydrodiscectomy (HydroD).

The purpose of this study is to compare the outcomes of HydroD with the SpineJet Hydrodiscectomy System to transforaminal epidural steroid injections (TESI) in patients with lumbar radiculopathy due to contained disc herniation that have failed a course of conservative management including anti-inflammatory medication and physical therapy. Patients will be randomized in a 1:1 ratio to Percutaneous Hydrodiscectomy or Transforaminal Epidural Steroid Injections.

Patients randomized to the TESI group that fail to have >50% relief of pain after two courses of TESI injections spaced two weeks apart within 2 months of the procedure, will be provided with the option to cross-over to the HydroD group after which they will follow the same follow-up visits. If after cross-over into the HydroD group they fail to have >50% relief of pain after the initial intervention within 2 months of the procedure, they will be referred for surgery and their participation in the study will end.

Patients randomized to the HydroD group that fail to have >50% relief of pain after the initial procedure, or within 2 months of the procedure, will be provided with the option to cross-over to the TESI group. If after cross-over to the TESI group they fail to have >50% relief of pain after two courses of TESI injections spaced two weeks apart within 2 months of the procedure, they will be referred for surgery and will no longer be followed in the study.

Patients will be followed at 1, and 4, and 2, 6, 12, and 24 months post-procedure. Outcomes assessments include NRS for pain, ODI, neurological and independent physician evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Single level subligamentous lumbar disc herniation with a size of up to 1/3 of the spinal canal sagittal diameter, with unilateral radicular pain attributed to nerve root impingement from lumbar disc material correlated with MRI or CT findings
* Axial MRI demonstrating unilateral focal contained disc herniation with single nerve contact
* Patient failed at least 3 weeks of conservative management within a 6 month period including anti-inflammatory medication and physical therapy
* Patient has not had previous epidural steroid injections at the affected lumbar level within 3 months of presenting for the study
* Patient is a candidate for transforaminal epidural steroid injections
* Positive Straight Leg Raising (SLR) test
* Patient has a leg pain > back pain
* The subject is physically and mentally able to participate in the study
* Patient is willing and able to provide informed consent
* Patient is willing and able to comply with the study protocol

Exclusion Criteria:

* Patient has had surgery at the affected level
* Extruded or sequestered disc herniation
* Free fragment herniation
* Discogenic pain without nerve root compression
* Previous surgery at the involved lumbar level
* Segmental instability (motion on flexion/extension films)
* Spondylolisthesis > Grade 2
* Severe central canal stenosis or bony impingement at the index level
* Significant loss of disc height (> 60%) compared with the adjacent higher level or disc height < 6mm at affected level
* Motor deficit (strength rating less than 4/5 in the lower extremity test)
* Positive Waddell test (> 3 of 5 tests)
* Active local or systemic infection
* Actively in litigation for pain symptoms
* Currently on Workman's Compensation
* Women who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed E Wahezi, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Hydrodiscectomy | TESI
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Hydrodiscectomy | TESI | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (5) | 45 (0) | 45 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Group That Experience at Least a 50% Reduction in Leg and Back Pain
Description: Pain improvement in all patients in HydroD arm with at least 50% reduction in leg and back pain.
Time Frame: 6 months
Population: Data were not collected.
Arm/Group | Percutaneous Hydrodiscectomy | TESI
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline Oswestry Disability Index (ODI)
Time Frame: 24 months
Population: Data were not collected
Arm/Group | Percutaneous Hydrodiscectomy | TESI
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline ED-5Q Questionnaire
Time Frame: 24 months
Population: Data were not collected
Arm/Group | Percutaneous Hydrodiscectomy | TESI
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Global Improvement Impression of Change (PGIC)
Description: Patient self assessment of the Global Improvement Impression of Change (PGIC)
Time Frame: 24 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Independent Physician Assessment (McNab Criteria)
Time Frame: 24 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Adverse Events
Description: Procedure and device related adverse events
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Percutaneous Hydrodiscectomy | TESI
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes